CLINICAL TRIAL: NCT00641173
Title: Early Intervention for PTSD in Iraqi Veterans
Brief Title: Early Intervention for Post Traumatic Stress Disorder (PTSD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn by funding source
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Bremner, Doug - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHBA-009-06F
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Post-Traumatic Stress Disorders
Keywords: PTSD; cortisol; hippocampus; memory
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): paroxetine v placebo
  Interventions: Drug: paroxetine
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: paroxetine — treatment with SSRI paroxetine
  Arms: 1
Drug: placebo — treatment with placebo
  Arms: 2

SUMMARY:
Over 150,000 soldiers are currently deployed in Iraq as part of Operation Iraqi Freedom (OIF), and 12% of returning OIF veterans have posttraumatic stress disorder (PTSD). Intervening soon after the trauma is critical for long-term outcomes, since with time traumatic memories become resistant to treatment. The current study will compare treatment with the selective serotonin reuptake inhibitor (SSRI) paroxetine to placebo in returning OIF veterans who have returned from Iraq in the past six months, who meet criteria for early PTSD. Assessment of PTSD symptoms, brain markers, neuropsychological testing of memory, and cortisol response to an Iraq-related traumatic script before and after the intervention are proposed to provide information about the effects of the interventions on PTSD symptoms and stress-responsive hormonal systems.

DETAILED DESCRIPTION:
Over 150,000 soldiers are currently deployed in Iraq as part of Operation Iraqi Freedom (OIF), and 12% of returning OIF veterans have posttraumatic stress disorder (PTSD). 389,100 soldiers developed chronic PTSD from the Vietnam War, requiring a life-time of VA mental health care. These veterans have suffered from a loss of work productivity, but also show greater utilization of health care resources and higher rates of physical disease. Research from our group and others showed lasting neurobiological consequences of PTSD, including an increased cortisol response to traumatic reminders, verbal declarative memory problems,6 and smaller hippocampal volume that reverses with treatment with the serotonin reuptake inhibitor (SSRI) paroxetine or the anticonvulsant phenytoin. Recently we found that three months of treatment with paroxetine in PTSD patients resulted in an increase in hippocampal N-acetyl-aspartate (NAA), a marker of neuronal integrity. Subjects treated with placebo did not have an increase in NAA, however subsequent treatment for three months with open label paroxetine resulted in an increase in NAA to the level seen in the subjects treated with paroxetine in the double-blind phase. Intervening soon after the trauma is critical for long-term outcomes, since with time traumatic memories become indelible and resistant to treatment. Diminished efficacy of treatment over time is shown by the fact that trials of Vietnam veterans have shown less efficacy over the years. Animal studies show that pretreatment before stress with antidepressants reduces chronic behavioral deficits related to stress; although for ethical and other reasons no studies have provided pretreatment before trauma exposure in humans. No studies have looked at the ability of antidepressants to treat early PTSD, which we are seeing in great numbers in veterans returning from OIF. This is important, since medications are not without side effects, and we cannot assume that early PTSD in Iraq veterans is the same as, for example, chronic Vietnam-related PTSD. Obtaining information about the risks and benefits of early treatment of PTSD in OIF veterans is critical to guiding treatment approaches to this emerging population. In addition, little is known about potential biomarkers of treatment response. We are working with the Georgia National Guard 48th Combat Brigade to evaluate the health needs of returning OIF veterans, and have started an OIF/OEF Trauma Clinic at the Atlanta VAMC where the PI is screening returning OIF veterans. We now propose to compare paroxetine and to placebo in returning OIF veterans who have returned from Iraq in the past six months, who meet criteria for early PTSD. Assessment of PTSD symptoms, hippocampal volume and NAA, neuropsychological testing of memory, and cortisol response to an Iraq-related traumatic script before and after the intervention are proposed to provide information about the effects of the interventions on PTSD symptoms and stress-responsive hormonal systems.

ELIGIBILITY:
Inclusion Criteria:

* Male and female veterans age 18-50
* Returned from Iraq Theater within the past six months
* Screen positive for PTSD related to Iraq deployment based on the PTSD Checklist
* Confirmed with PTSD based on the CAPS, including one month duration of symptoms
* Being discharged from active service from Iraq
* Provide written informed consent

Exclusion Criteria:

* History of loss of consciousness of more than one minute
* Psychotropic medication use within the previous four weeks
* History (based on the SCID) of lifetime or current alcohol or substance abuse/dependence, schizophrenia, schizoaffective disorder, or bipolar disorder.
* Positive urine toxicology screen
* History of pre-deployment-related PTSD or partial PTSD based on the CAPS
* History of PTSD or partial PTSD related to a prior deployment
* Serious medical or neurological illness
* Pregnancy
* History of asthma
* Steroid usage, both inhaled and oral
* Seizure disorder
* Prenatal/perinatal substance exposure or trauma.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
CAPS | three months

SECONDARY OUTCOMES:
hippocampal volume and NAA | three months
memory | three months
cortisol response to stress | three months

CONTACTS AND LOCATIONS:
Overall Officials: Doug Bremner, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur